CLINICAL TRIAL: NCT06465004
Title: Exploratory Pilot Trial Assessing the Immediate Impact of Animal-based and Plant-based Protein Drinks on Blood Parameters
Brief Title: Pilot Trial: Bioavailability Animal vs. Plant Protein Drink
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-00151
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Nutrition, Healthy; Leucine Sensitivity
Keywords: Leucin; Plant-based; Animal-based; Bioavailability

STUDY DESIGN:
Intervention Model Description: Randomized cross-over design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Animal-based A (Active Comparator): A commercially available high protein drink, based on animal proteins (Fresubin Protein Energy)
  Interventions: Dietary Supplement: Consumption of protein - rich drink
- Animal-based B (Active Comparator): A homemade drink containing animal-based proteins, using a specific animal-based protein isolate mix.
  Interventions: Dietary Supplement: Consumption of protein - rich drink
- Plant-based A (Active Comparator): A homemade drink containing plant-based proteins, formulated to have the same macronutrient content as the animal-based drinks.
  Interventions: Dietary Supplement: Consumption of protein - rich drink

INTERVENTIONS:
Dietary Supplement: Consumption of protein - rich drink — The participants will drink on of three protein - rich drinks

SUMMARY:
A pilot study is being conducted to compare a new plant-based protein drink to commercially available animal-based protein drinks. The goal is to assess if the plant-based drink delivers amino acids to the bloodstream as effectively as the animal-based drinks, potentially offering a viable option for those on plant-based diets.

The study will involve approximately 12 healthy adults aged 18-40. Each participant will try all three drinks (the new plant-based drink, a commercial animal-based drink, and another animal-based recipe) on separate days in a randomized order. Before and after (30, 60, and 90 minutes) consuming each drink, a small blood sample will be drawn to measure amino acid levels (leucine).

By comparing the results, the investigators hope to determine if the plant-based drink can match the effectiveness of animal-based protein drinks in delivering essential nutrients. This research could contribute to the development of sustainable and nutritious plant-based protein alternatives.

ELIGIBILITY:
Inclusion criteria

* Gender: male and female
* Age: 18-40 years
* Signed written informed consent

Exclusion criteria

* Smoking history
* Cardiovascular diseases
* BMI > 35 kg/m2
* Caffeine consumption < 1 day before the study participation
* Allergies: Soy, Peas, Milk, Lactose, Fructose
* High intensity exercise <2 days before study participation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-06-08 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
leucine content in the blood | 4 hours
  Assessment of leucine content in blood before and 30-60-90 min after consumption of drink

CONTACTS AND LOCATIONS:
Overall Officials: Gommaar D'Hulst, PhD, Principal Investigator — ETH Zurich
Locations (1):
- SLA - ETH Zurich, Schwerzenbach, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/04/NCT06465004/Prot_SAP_000.pdf